CLINICAL TRIAL: NCT03457181
Title: Effect of Music on Patient's Anxiety, Satisfaction and Pain During Carotid Endarterectomy: Multicenter Prospective Randomized Controlled Trial
Brief Title: Effect of Music During Carotid Endarterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AntalyaTRH 19
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Active Comparator): in music group, patient was asked to choose one music genres from 5 different music genres according to his/her preference. Patient selected music was delivered by an iPhone 6 and Music app (Apple Inc., USA) through the iPhone's headphones.
  Interventions: Other: music
- operating room noise group (Active Comparator): in operating room noise group, operating room noise was delivered by an iPhone and Microphone App (Free version, Von Bruno). This application allows the iPhone to be used as a live microphone.
  Interventions: Other: operating room noise

INTERVENTIONS:
Other: music — effect of music on anxiety scores
  Arms: music group
Other: operating room noise — effect of operating room noise on anxiety scores
  Arms: operating room noise group

SUMMARY:
The purpose of this study is to test the hypothesis that music listening during carotid endarterectomy administered the cervical plexus block will cause less anxiety, less pain, and greater patient satisfaction.

DETAILED DESCRIPTION:
Patients who decided to participate in the study were randomized by means of a computer-generated randomization order into 2 groups: Music Group (Group M) and Operating Room (OR) Noise Group (Group O). Randomization was independently carried out in both centers.

Preoperative and postoperative State Trait Anxiety Inventory (STAI) scores, intraoperative STAI responses, preoperative and postoperative numerical rating scale scores for anxiety, pain scores and hemodynamic parameters were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing carotid endarterectomy using cervical plexus block
* American Society of Anesthesiologists class 2 to 3
* Ability to consent

Exclusion Criteria:

* inability to communicate
* not understand the aim and objectives of the study
* not provide informed written consent
* contraindications for the block (local infection, coagulation disorders)
* hypersensitivity to the local anesthetics
* refusal of regional anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Differences in intraoperative State-Trait Anxiety Inventory Response (relaxed ) | 60 minutes
  Assessed every 5 minutes during the procedure. The question is "are you relaxed" and patient is asked to answer the question on a scale of "very much, moderately, somewhat, or not at all"

SECONDARY OUTCOMES:
Differences in intraoperative State-Trait Anxiety Inventory Response (calm) | 60 minutes
  Assessed every 5 minutes during the procedure. The questions is "are you calm" and patient is asked to answer the question on a scale of "very much, moderately, somewhat, or not at all"
Differences in postoperative anxiety numerical rating scale scores | 10 minutes
  assessed 5 min after the procedure. Numeric Rating Scale (NRS): from 0 (no anxiety) to 10 (worst feeling of anxiety possible)
Differences in preoperative State-Trait Anxiety Inventory scores | 20 minutes
  assessed 1 day before surgery. The total score on the scale ranges from 20 to 80 points and a higher score represents greater anxiety.
Differences in postoperative State-Trait Anxiety Inventory scores | 20 minutes
  assessed 1st day after surgery. The total score on the scale ranges from 20 to 80 points and a higher score represents greater anxiety.
Differences in pain scores | 10 minutes
  assessed 5th min after surgery. (from 0 (no pain) to 10 (maximal possible pain))
Changes in mean arterial pressure | 60 minutes
  Assessed every 5 minutes during the procedure
Changes in heart rate | 60 minutes
  Assessed every 5 minutes during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, M.D., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research hospital, Antalya, Turkey (Türkiye)